CLINICAL TRIAL: NCT02502942
Title: Effects of Upper Airway Muscle Training on Obstructive Sleep Apnea (OSA)
Brief Title: Effects of Upper Airway Muscle Training on OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Robert L. Owens, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: UCSD130780; R01HL085188-05A1 (NIH)
Record Dates: First submitted 2015-07-12; First posted 2015-07-20 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Exercise; Upper airway muscle
MeSH Terms: conditions — Sleep Apnea, Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Untreated OSA Muscle Exercise Group (Experimental): Patients who were previously diagnosed of obstructive sleep apnea (OSA) with apnea hypopnea index (AHI) > 10 events/hr and have previously failed or refused PAP therapy. In this group, patients will learn and practice upper airway muscle exercise for six weeks.
  Interventions: Behavioral: Upper Airway Muscle Exercise
- PAP Therapy Muscle Exercise Group (Experimental): OSA patients who are currently treated with PAP for their OSA (with AHI of previous sleep study > 10 events/hr). In this group, patients will learn and practice upper airway muscle exercise for six weeks.
  Interventions: Behavioral: Upper Airway Muscle Exercise
- Oral Appliance Muscle Exercise Group (Experimental): OSA patients who are currently treated with an oral appliance with residual AHI > 10 events/hr. In this group, patients will learn and practice upper airway muscle exercise for six weeks.
  Interventions: Behavioral: Upper Airway Muscle Exercise
- Normal Control Sham Exercise Group (Active Comparator): Patients of untreated OSA group, PAP therapy group, and oral appliance group are randomized to upper airway muscle exercise versus sham exercise.
  Interventions: Behavioral: Sham Exercise

INTERVENTIONS:
Behavioral: Upper Airway Muscle Exercise — Patients will use an individualized oral retainer device for upper airway muscle training exercises daily for 20 minutes each day (10 minutes in the morning and 10 minutes in the afternoon/evening) for 6 weeks.
  Arms: Oral Appliance Muscle Exercise Group; PAP Therapy Muscle Exercise Group; Untreated OSA Muscle Exercise Group
Behavioral: Sham Exercise — Patients will be given an individualized oral retainer device and instructed to do deep breathing exercise twice daily for 6 weeks.
  Arms: Normal Control Sham Exercise Group

SUMMARY:
Obstructive sleep apnea (OSA) is a common disorder characterized by recurrent collapse of the upper airway during sleep. OSA patients have a small upper airway that is kept patent during wakefulness by a compensatory increase in upper airway (UA) dilator muscle (e.g. genioglossus) activity. At sleep onset this compensation is reduced or lost, resulting in upper airway narrowing or collapse. Previous studies of upper airway muscle training showed variable results on OSA, but so far there has not been any practical, long-term, systematic upper airway muscle training developed or studied as the treatment of OSA. In theory, strengthening the upper airway muscle with exercise training in theory helps maintain a patent airway during sleep. Therefore, investigators aim to test the hypothesis: 1) UA muscle training can improve sleep apnea in some patients with OSA, including those already receiving treatment with PAP or oral appliance therapy. 2) Muscle training is a viable therapy for a definable subset of OSA patients. Investigators hypothesize that patients with OSA who have mild or moderately compromised upper airway anatomy will benefit the most. 3)There will be a positive association between the changes in muscle function and improvement in OSA severity.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common disorder characterized by recurrent collapse of the upper airway during sleep, which leads to recurrent arousal and subsequent daytime sleepiness. The most commonly accepted reason for the initiation of obstructive respiratory events in OSA is that patients have a small upper airway that is kept patent during wakefulness by a compensatory increase in upper airway dilator muscle (e.g. genioglossus) activity. At sleep onset this compensation is reduced or lost, resulting in upper airway narrowing or collapse.

Upper airway (UA) muscle training appears to have some benefit in OSA with improvement in the AHI, although the current data shows variable results, particularly when publication bias is taken into account. Many remain skeptical about these data based on clinical experience and prior negative studies (which remain largely unpublished). Moreover, previous positive studies involved exercises that are usually impractical to be continued in the long-term.

Therefore, investigators will undertake a rigorous assessment of a practical UA muscle training on OSA. Investigators will recruit patients with OSA that are wither unable/unwilling to use CPAP, as well as those who are already on treatment with PAP or oral appliances. The exercises include 4 steps: step 1 is to put on an individualized fitted oral retainer device to guide the exercise; step 2 is to push the tongue towards the hard palate to press the movable part of the oral retainer device for 4 minutes; step 3 is to touch the hard palate using the middle part of the tongue, hold for 10 seconds and repeat it for 4 minutes; step 4 is to remove the retainer device and brush the tongue gently on both sides for 2 minute. The exercise will take 20 minutes a day (10 minutes in the morning and 10 minutes in the afternoon/evening).

Investigators will study the effect of upper airway (UA) muscle training on OSA severity, muscle strengh and endurance. Investigators aim to determine the characteristics of OSA patients most likely to benefit from UA muscle training and the association between changes in muscle function and OSA severity.

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis of OSA with AHI>10 events/hr.
* PAP group: subjects who have been on PAP treatment for at least 3 month, with good compliance (at least 4 hours a day and use PAP for >70% of the time).
* Untreated group: untreated subjects with generally mild OSA as defined by AHI<20 events/hr and nadir SaO2>70%. Additionally, investigators will also recruit OSA subjects of all severities who have previously tried but are not currently using PAP.
* Oral appliance treatment group: subjects have residual AHI >10 events/hr with oral appliance therapy.

Exclusion Criteria:

* In those with untreated sleep apnea, severe sleepiness with current Epworth Sleepiness Scale (ESS) > 18 or history of motor vehicle accident due to obstructive sleep apnea
* Taking medications classified as a muscle relaxant
* Pregnant women.
* Psychiatric disorder, other than mild and controlled depression; e.g. schizophrenia, bipolar disorder, major depression, panic or anxiety disorders.
* Current smokers, alcohol (>3oz/day) or use of illicit drugs.
* More than 10 cups of beverages with caffeine (coffee, tea, soda/pop) per day.
* Unstable cardiac disease (e.g. congestive heart failure)
* Pulmonary disease (apart from well controlled mild asthma and OSA)
* Systemic neuromuscular disease
* Other systemic disease that affects breathing (e.g. stroke) or those with expected survival < 1 year.
* Poor oral condition, including: active periodontal disease, loose or broken teeth, lack of eight teeth in each arch, active TMJ dysfunction
* Known allergy to oral appliance components

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2015-08; Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
Change of severity of obstructive sleep apnea, measured as apnea hypopnea index (AHI), for untreated OSA group and oral appliance group | Baseline and after 6-week exercise training
  Home sleep test is used to measure AHI.
Change of severity of obstructive sleep apnea, measured as 95th percentile pressures, for PAP therapy group | Baseline and after 6-week exercise training
  95th percentile pressures (2 week period) of autotitrating CPAP will be used to assess the effects of upper airway muscle exercise on muscle strength.

SECONDARY OUTCOMES:
Change of sleepiness measured by Epworth Sleepiness Scale (ESS) | Baseline and after 6-week exercise training
  ESS is a self-administered questionnaire with 8 questions. It provides a measure of a person's general level of daytime sleepiness, or their average sleep propensity in daily life.
Change of sleep quality measured by Pittsburgh Sleep Quality Index (PSQI) | Baseline and after 6-week exercise training
  PSQI is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval.
Change of subjective quality of life measured by SF-36 | Baseline and after 6-week exercise training
  SF-36 is a patient-reported survey of patient health status.
Change of neurocognitive function measured by psychomotor vigilance test (PVT) | Baseline and after 6-week exercise training
  PVT is a sustained-attention, reaction-timed task that measures the speed with which subjects respond to a visual stimulus.
Change of upper airway anatomy evaluated with acoustic pharyngometry | Baseline and after 6-week exercise training
  Acoustic pharyngometry is a non-invasive sonic measurement of the upper airway anatomy.
Change of tongue strength and endurance evaluated with Iowa Oral Performance Instrument (IOPI) | Baseline and after 6-week exercise training
  IOPI is a hand held manometer which measures intraoral pressure generated by compression of an air filled bulb by the tongue against the palate.

CONTACTS AND LOCATIONS:
Overall Officials: Atul Malhotra, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States